CLINICAL TRIAL: NCT04507087
Title: Randomized Controlled Trial of a Documentary to Encourage Plant-based Eating
Brief Title: Documentary to Encourage Plant-based Eating
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Maya Mathur, Assistant Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: eatingveg
Record Dates: First submitted 2020-07-31; First posted 2020-08-11 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Eating Behavior
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): See detailed preregistration: https://osf.io/xrckh/registrations
  Interventions: Behavioral: Documentary
- Control (Sham Comparator): See detailed preregistration: https://osf.io/xrckh/registrations
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Documentary — A 20-minute documentary about the health, environmental, and animal welfare consequences of eating meat and animal products
  Arms: Intervention
Behavioral: Control — A 20-minute unrelated video (a motivational talk entitled "Listening to shame")
  Arms: Control

SUMMARY:
This study will assess whether watching a documentary video about the health, environmental, and ethical consequences of eating meat and animal products reduces participants' self-reported intake of these items.

DETAILED DESCRIPTION:
See detailed preregistration: https://osf.io/xrckh/registrations

ELIGIBILITY:
Inclusion Criteria:

* Participant is currently located in the United States
* Participant is at least 18 years old

Exclusion Criteria:

* Participant is located outside the United States
* Participant is less than 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 650 (Actual)
Dates: Start 2020-08-26 (Actual); Primary Completion 2020-09-07 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Total meat and animal product consumption | Consumption over the 1-week time frame spanning approximately 1 week to 2 weeks after baseline data collection
  Self-reported meat and animal product consumption (ounces consumed over the past week)

SECONDARY OUTCOMES:
Total meat consumption | Consumption over the 1-week time frame spanning approximately 1 week to 2 weeks after baseline data collection
  Self-reported meat consumption (ounces consumed over the past week)
Total animal product consumption | Consumption over the 1-week time frame spanning approximately 1 week to 2 weeks after baseline data collection
  Self-reported animal product consumption (ounces consumed over the past week)
Consumption of each of 8 individual categories of meats and animal products | Consumption over the 1-week time frame spanning approximately 1 week to 2 weeks after baseline data collection
  Self-reported consumption (ounces consumed over the past week)
Total consumption of selected, healthy plant-based foods (ounces consumed over the past week) | Consumption over the 1-week time frame spanning approximately 1 week to 2 weeks after baseline data collection
  Self-reported consumption (ounces consumed over the past week)

OTHER OUTCOMES:
Perceived importance of health | 2 weeks after baseline data collection
  A single Likert item adapted from Heckler (2010), ranging from 1 to 6, with higher scores representing greater perceived importance. The exact text is provided in detailed preregistration: https://osf.io/xrckh/registrations.
Perceived importance of environmental sustainability | 2 weeks after baseline data collection
  A single Likert item adapted from Heckler (2010), ranging from 1 to 6, with higher scores representing greater perceived importance. The exact text is provided in detailed preregistration: https://osf.io/xrckh/registrations.
Perceived importance of animal welfare | 2 weeks after baseline data collection
  A single Likert item adapted from Heckler (2010), ranging from 1 to 6, with higher scores representing greater perceived importance. The exact text is provided in detailed preregistration: https://osf.io/xrckh/registrations.
Speciesism | 2 weeks after baseline data collection
  Caviola et al.'s (2019) Speciesism Scale, consisting of 6 Likert items each ranging from 1 to 7. After reverse-coding, a higher score on the sum of the items (ranging from 6 to 42) represents greater speciesism. The exact text for all items is provided in detailed preregistration: https://osf.io/xrckh/registrations.
Interest in animal welfare activism and reform | 2 weeks after baseline data collection
  2 items modified from Corning et al.'s (2002) Activism Orientation Scale as well as 3 novel items, consisting in total of 5 items each ranging from 1 to 7. A higher score on the sum of the items (ranging from 5 to 35) represents greater interest in activism and reform. The exact text for all items is provided in detailed preregistration: https://osf.io/xrckh/registrations.
Social dominance orientation | 2 weeks after baseline data collection
  Ho et al.'s (2015) 8-item Social Dominance Orientation [SDO(7)] scale, consisting in total of 5 items each ranging from 1 to 7. After reverse-coding, a higher score on the sum of the items (ranging from 8 to 56) represents greater interest in activism and reform. The exact text for all items is provided in detailed preregistration: https://osf.io/xrckh/registrations.

CONTACTS AND LOCATIONS:
Overall Officials: Maya B Mathur, PhD, Principal Investigator — Stanford University
Locations (1):
- Maya Mathur, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: Yes
All materials and analysis code required to reproduce all results will be made publicly available. All data except for participants' counties of residence (which is considered identifying information) will also be made publicly available.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Immediately upon journal acceptance or earlier if possible given embargo policies.
Access Criteria: Public availability
URL: https://osf.io/xrckh/

REFERENCES:
- See also: Future location of data, code, and materials — https://osf.io/xrckh/
- See also: Detailed preregistration — https://osf.io/xrckh/registrations